CLINICAL TRIAL: NCT03535337
Title: Adaptive Antiretroviral Therapy Adherence Interventions for Youth Living With HIV Through Text Messaging and Cell Phone Support Embedded Within the Sequential Multiple Assignment Randomized Trial (SMART) Design
Brief Title: Adherence Interventions for HIV Youth Via Text & Cell Phone - Sequential Multiple Assignment Randomized Trial (SMART)
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Children's Hospital Los Angeles (Other); Hunter College of City University of New York (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Sylvie Naar, Principal Investigator, Florida State University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ATN 144
Record Dates: First submitted 2018-04-12; First posted 2018-05-24 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: Interventions; youth living with HIV; mHealth; ART adherence; adaptive intervention; cell phone; text messaging
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Multiple Assignment Randomized Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- CPS-Rsp-T (Active Comparator): After 3 months of intervention, this group of CPS Rsp will receive 3 months of CPS-T intervention followed by SC.
  Interventions: Behavioral: CPS
- CPS-Rsp-SC (Active Comparator): After 3 months of intervention, this group of CPS Rsp's intervention will discontinue and they'll receive SC only
  Interventions: Behavioral: CPS
- CPS-NRsp-I (Active Comparator): After 3 months of intervention, this group of CPS NRsp will receive 3 months of CPS-I followed by 3 months of CPS-T and 3 months of SC.
  Interventions: Behavioral: CPS
- CPS-NRsp-SMS-I (Active Comparator): After 3 months of intervention, this group of CPS NRsp will receive 3 months of SMS-I followed by 3 months of SMS-T and 3 months of SC
  Interventions: Behavioral: CPS
- SMS-Rsp-T (Active Comparator): After 3 months of intervention, this group of SMS Rsp will receive 3 months of SMS tapered (SMS-T) intervention followed by SC.
  Interventions: Behavioral: SMS
- SMS-Rsp-SC (Active Comparator): After 3 months of intervention, this group of SMS Rsp, intervention will discontinue and they'll receive SC only
  Interventions: Behavioral: SMS
- SMS-NRsp-CPS-I (Active Comparator): After 3 months of intervention, this group of SMS NRsp will receive 3 months of CPS-I followed by 3 months CPS-T and 3 months SC
  Interventions: Behavioral: SMS
- SMS-NRsp-I (Active Comparator): After 3 months of intervention, this group of SMS NRsp will receive 3 months of SMS-I followed by 3 months of SMS-T and 3 months of SC
  Interventions: Behavioral: SMS

INTERVENTIONS:
Behavioral: CPS — Assessment of participant's medication adherence and barrier problem solving via phone conversation
  Arms: CPS-NRsp-I; CPS-NRsp-SMS-I; CPS-Rsp-SC; CPS-Rsp-T
Behavioral: SMS — Participants will receive a text message, which will be an electronic reminder regarding medication adherence. Participants will then text back a confirmatory response.
  Arms: SMS-NRsp-CPS-I; SMS-NRsp-I; SMS-Rsp-SC; SMS-Rsp-T

SUMMARY:
The purpose of this study is to test an adaptive adherence intervention, which utilizes two mobile health (mHealth) intervention designs, in an effort to promote adherence to antiretroviral therapy (ART) and achieve and maintain viral load (VL) suppression in youth living with HIV (YLH) while increasing understanding of the context for wide-scale implementation of cell phone support (CPS) and text messaging support (SMS), with and without incentives.

DETAILED DESCRIPTION:
The study will consist of two points of randomization. The first step involves randomization of participants to receive either CPS or SMS using a 1:1 allocation ratio. Both intervention conditions will receive 3 months of intervention (i.e., 12 weeks of CPS or SMS).

The second step involves a stratified randomization in blocks with 8 possible intervention trajectories. Within each condition, participants are categorized into two groups - responders with VL<200 (Rsp) and non-responders with VL ≥200 (NRsp). Responders in the CPS condition will be randomly assigned to receive either 3 months of CPS tapered (CPS-T) intervention followed by standard care (SC) or only SC. Similarly, responders in the SMScondition will be randomly assigned to receive either 3 months of SMS tapered (SMS-T) intervention followed by SC or only SC. Non-responders in both CPS and SMS conditions will be randomly assigned to receive either 3 months of incentivized CPS (CPS-I) followed by 3 months of CPS-T and 3 months of SC or 3 months of incentivized SMS (SMS-I) followed by 3 months of SMS-T and 3 months of SC.

ELIGIBILITY:
Inclusion Criteria:

* HIV diagnosis
* Viral load ≥ 200 copies/mL within 3 months prior to enrollment or self-reported adherence ≤ 80%
* ART medication regimen prescribed minimum of 3 months prior to eligibility VL or self-reported adherence
* Sole owner of device capable of sending/receiving calls and text messages
* Willingness to permit research team to communicate with their HIV care provider team

Exclusion Criteria:

* Mental, physical, or emotional capacity prevents completion of protocol as written
* Inability to understand written/spoken English
* Concurrent participant in any adherence behavioral research intervention

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The City University of New York, New York, New York, United States

REFERENCES:
- [Derived] Belzer ME, MacDonell KK, Ghosh S, Naar S, McAvoy-Banerjea J, Gurung S, Cain D, Fan CA, Parsons JT. Adaptive Antiretroviral Therapy Adherence Interventions for Youth Living With HIV Through Text Message and Cell Phone Support With and Without Incentives: Protocol for a Sequential Multiple Assignment Randomized Trial (SMART). JMIR Res Protoc. 2018 Dec 20;7(12):e11183. doi: 10.2196/11183. PMID 30573448

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1 Cell Phone Support: CPS: Assessment of participant's medication adherence and barrier problem solving via phone conversation
- Stage 1 Short Message Service (SMS): SMS: Participants will receive a text message, which will be an electronic reminder regarding medication adherence. Participants will then text back a confirmatory response.
- Stage 2 Cell Phone Support CPS-I: Cell Phone Support Non-responder re-randomized to cell phone support incentivized
- Stage 2 Cell Phone Support SMS-I: Cell phone support non-responder, re-randomized to SMS incentivized
- Stage 2 Cell Phone Support CPS-T: Cell phone support responder, re-randomized to cell phone support tapered
- Stage 2 Cell Phone Support SC: Cell phone support responder, re-randomized to standard of care
- Stage 2 Short Message Service SMS-T: Short message service (SMS) responder, re-randomized to SMS tapered
- Stage 2 Short Message Service SC: Short message service responder, re-randomized to standard of care
- Stage 2 Short Message Service CPS-I: Short message service non-responder, re-randomized to cell phone support incentivized
- Stage 2 Short Message Service SMS-I: Short message service non-responder, re-randomized to SMS incentivized
Period: Stage 1 Randomization
Arm/Group | Stage 1 Cell Phone Support | Stage 1 Short Message Service (SMS) | Stage 2 Cell Phone Support CPS-I | Stage 2 Cell Phone Support SMS-I | Stage 2 Cell Phone Support CPS-T | Stage 2 Cell Phone Support SC | Stage 2 Short Message Service SMS-T | Stage 2 Short Message Service SC | Stage 2 Short Message Service CPS-I | Stage 2 Short Message Service SMS-I
Started | 40 | 43 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 40 | 43 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2 Randomization
Arm/Group | Stage 1 Cell Phone Support | Stage 1 Short Message Service (SMS) | Stage 2 Cell Phone Support CPS-I | Stage 2 Cell Phone Support SMS-I | Stage 2 Cell Phone Support CPS-T | Stage 2 Cell Phone Support SC | Stage 2 Short Message Service SMS-T | Stage 2 Short Message Service SC | Stage 2 Short Message Service CPS-I | Stage 2 Short Message Service SMS-I
Started | 0 | 0 | 2 | 4 | 11 | 16 | 14 | 14 | 3 | 5
Completed | 0 | 0 | 0 | 3 | 6 | 12 | 11 | 8 | 3 | 3
Not Completed | 0 | 0 | 2 | 1 | 5 | 4 | 3 | 6 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1 | 5 | 4 | 3 | 6 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Cell Phone Support | Stage 1 Short Message Service (SMS) | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.58 (1.63) | 21.9 (1.80) | 22.27 (1.78)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 32 | 35 | 67
  Female | 5 | 6 | 11
  Other | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 20 | 24 | 44
  Latino | 9 | 10 | 19
  White | 4 | 3 | 7
  Multiracial/Other | 7 | 6 | 13
Region [Count of Participants; unit: Participants]
  Northeast United States | 3 | 8 | 11
  Midwest United Stated | 8 | 4 | 12
  Southeastern United States | 20 | 24 | 44
  Western United States | 9 | 7 | 16
Employed [Count of Participants; unit: Participants] | 24 | 20 | 44
Education [Count of Participants; unit: Participants]
  Less than High School | 7 | 6 | 13
  High School or Equivalent | 17 | 15 | 32
  Some College or Above | 16 | 22 | 38
Sexual Identity [Count of Participants; unit: Participants]
  Gay | 29 | 34 | 63
  Heterosexual or Other | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Undetectable Viral Load
Description: Percent of participants that have an undetectable HIV Viral Load.
Time Frame: baseline, month 3, month 6, month 9, and month 12
Population: Significant attrition at follow-ups for viral load testing. Therefore the overall model would not converge.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1 Cell Phone Support | Stage 1 Short Message Service (SMS) | Stage 2 Cell Phone Support CPS-I | Stage 2 Cell Phone Support SMS-I | Stage 2 Cell Phone Support CPS-T | Stage 2 Cell Phone Support SC | Stage 2 Short Message Service SMS-T | Stage 2 Short Message Service SC | Stage 2 Short Message Service CPS-I | Stage 2 Short Message Service SMS-I
Number analyzed (Participants) | 34 | 35 | 1 | 1 | 7 | 8 | 9 | 12 | 1 | 2
percentage of participants
  Baseline: number analyzed (Participants) | 34 | 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline | 58.8 | 62.9 |  |  |  |  |  |  |  |
  3 Month: number analyzed (Participants) | 19 | 24 | 1 | 1 | 6 | 8 | 9 | 12 | 0 | 0
  3 Month | 89.5 | 87.5 | 100 | 100 | 100 | 100 | 90.0 | 100 |  |
  6 Month: number analyzed (Participants) | 16 | 19 | 1 | 0 | 6 | 6 | 8 | 6 | 0 | 2
  6 Month | 93.8 | 89.5 | 100 |  | 85.7 | 100 | 100 | 85.7 |  | 100
  9 Month: number analyzed (Participants) | 12 | 12 | 1 | 1 | 4 | 4 | 4 | 5 | 0 | 1
  9 Month | 83.3 | 83.3 | 100 | 100 | 80.0 | 80.0 | 100 | 83 |  | 100
  12 Month: number analyzed (Participants) | 5 | 6 | 0 | 0 | 3 | 2 | 3 | 1 | 1 | 0
  12 Month | 80.0 | 100.0 |  |  | 100 | 50.0 | 100 | 100 | 100 |

2. Primary Outcome: Medication Adherence Rate - 7 Day
Description: Self reported percentage of medication taken in the past 7 days prior to assessment point. Medication adherence rates will be compared between CPS and SMS groups.
Time Frame: baseline, month 3, month 6, month 9, and month 12
Population: Numbers are different due to attrition.
Measure: Mean (Standard Deviation); unit: percentage of medication adherence
Groups:
- Stage 2: Cell Phone Support CPS-I: Cell Phone Support non-responder, re-randomized to cell phone support incentivized
- Stage 2 Short Message Service SMS-T: Short message service responder, re-randomized to SMS tapered
Arm/Group | Stage 1 Cell Phone Support | Stage 1 Short Message Service (SMS) | Stage 2: Cell Phone Support CPS-I | Stage 2 Cell Phone Support SMS-I | Stage 2 Cell Phone Support CPS-T | Stage 2 Cell Phone Support SC | Stage 2 Short Message Service SMS-T | Stage 2 Short Message Service SC | Stage 2 Short Message Service CPS-I | Stage 2 Short Message Service SMS-I
Number analyzed (Participants) | 40 | 43 | 2 | 4 | 11 | 15 | 14 | 14 | 3 | 5
percentage of medication adherence
  Baseline: number analyzed (Participants) | 40 | 43 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline | 63.68 (34.91) | 74.52 (29.81) |  |  |  |  |  |  |  |
  3 month: number analyzed (Participants) | 39 | 34 | 1 | 2 | 11 | 15 | 13 | 14 | 2 | 5
  3 month | 90.69 (15.57) | 76.18 (34.20) | 70.00 (0.00) | 100 (0.00) | 94.60 (8.20) | 88.00 (19.30) | 95.40 (8.80) | 79.30 (32.50) | 15.00 (21.20) | 42.00 (35.60)
  6 month: number analyzed (Participants) | 22 | 32 | 2 | 3 | 8 | 9 | 13 | 12 | 2 | 5
  6 month | 80.00 (31.93) | 84.55 (20.09) | 100 (0.00) | 40 (45.80) | 96.30 (7.40) | 74.40 (33.20) | 94.60 (8.80) | 76.70 (28.10) | 95.00 (7.10) | 70.00 (24.50)
  9 month: number analyzed (Participants) | 22 | 36 | 2 | 3 | 7 | 10 | 11 | 8 | 3 | 5
  9 month | 79.17 (29.18) | 82.76 (23.89) | 100 (0.00) | 76.70 (40.40) | 85.70 (21.50) | 72.00 (35.50) | 94.60 (5.20) | 92.50 (7.10) | 56.70 (40.40) | 54.00 (28.80)
  12 month: number analyzed (Participants) | 19 | 24 | 0 | 3 | 5 | 11 | 10 | 8 | 3 | 3
  12 month | 73.33 (38.12) | 79.63 (30.19) |  | 33.30 (57.70) | 98.00 (4.50) | 79.10 (29.50) | 97.00 (6.70) | 70.00 (36.30) | 66.70 (25.20) | 46.70 (47.30)
Statistical Analysis 1: Comparison: Stage 1 Cell Phone Support vs Stage 1 Short Message Service (SMS); Test type: Superiority; p = 0.03, Mixed Models Analysis; Slope = 2.44, 95% CI 2-sided [0.28 to 4.59], Standard Error of Mean 1.10

3. Primary Outcome: Medication Adherence - 30 Days
Description: Self reported percentage of medication taken in the past 30 days prior to assessment point. Medication adherence rates will be compared between CPS and SMS groups.
Time Frame: baseline, month 3, month 6, month 9, and month 12
Population: Numbers are different due to attrition.
Measure: Mean (Standard Deviation); unit: percentage of medication adherence
Groups:
- Stage 2 Cell Phone Support CPS-I: Cell Phone Support non-responder, re-randomized to cell phone support incentivized
Arm/Group | Stage 1 Cell Phone Support | Stage 1 Short Message Service (SMS) | Stage 2 Cell Phone Support CPS-I | Stage 2 Cell Phone Support SMS-I | Stage 2 Cell Phone Support CPS-T | Stage 2 Cell Phone Support SC | Stage 2 Short Message Service SMS-T | Stage 2 Short Message Service SC | Stage 2 Short Message Service CPS-I | Stage 2 Short Message Service SMS-I
Number analyzed (Participants) | 31 | 36 | 2 | 2 | 10 | 14 | 13 | 13 | 3 | 4
percentage of medication adherence
  Baseline: number analyzed (Participants) | 31 | 36 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline | 68.55 (27.18) | 74.33 (23.60) |  |  |  |  |  |  |  |
  3 Month: number analyzed (Participants) | 27 | 30 | 1 | 2 | 10 | 14 | 12 | 13 | 1 | 4
  3 Month | 87.56 (20.35) | 84.87 (22.73) | 75.00 (0.00) | 53.00 (32.50) | 95.10 (6.00) | 88.00 (22.00) | 96.20 (4.60) | 83.90 (24.50) | 70.00 (0.00) | 58.00 (31.10)
  6 Month: number analyzed (Participants) | 21 | 31 | 2 | 2 | 8 | 9 | 13 | 11 | 2 | 4
  6 Month | 85.48 (21.14) | 82.13 (20.08) | 77.50 (23.30) | 88.50 (16.30) | 96.00 (9.80) | 77.20 (27.00) | 94.30 (8.40) | 73.50 (28.30) | 95.00 (7.10) | 55.00 (35.20)
  9 Month: number analyzed (Participants) | 23 | 27 | 2 | 2 | 7 | 10 | 11 | 7 | 3 | 4
  9 Month | 78.34 (27.92) | 83.74 (21.33) | 93.00 (1.40) | 90.50 (13.40) | 87.40 (21.70) | 67.90 (35.50) | 94.60 (6.00) | 91.10 (8.70) | 56.00 (39.30) | 58.00 (19.60)
  12 Month: number analyzed (Participants) | 18 | 25 | 0 | 2 | 5 | 10 | 10 | 7 | 3 | 2
  12 Month | 83.94 (22.73) | 80.60 (28.73) |  | 52.00 (67.90) | 94.00 (5.50) | 85.60 (12.80) | 97.10 (6.30) | 75.40 (29.80) | 69.00 (28.60) | 17.00 (24.00)
Statistical Analysis 1: Comparison: Stage 1 Cell Phone Support vs Stage 1 Short Message Service (SMS); Test type: Superiority; p = 0.82, Mixed Models Analysis; Slope = 0.17, 95% CI 2-sided [-1.32 to 1.66], Standard Error of Mean 0.76

ADVERSE EVENTS:
Time Frame: Every 1 Year, for up to 3 years and 9 months.
Arm/Group | Stage 1 Cell Phone Support | Stage 1 Short Message Service (SMS) | Stage 2 Cell Phone Support CPS-I | Stage 2 Cell Phone Support SMS-I | Stage 2 Cell Phone Support CPS-T | Stage 2 Cell Phone Support SC | Stage 2 Short Message Service SMS-T | Stage 2 Short Message Service SC | Stage 2 Short Message Service CPS-I | Stage 2 Short Message Service SMS-I
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43 | 0/2 | 0/4 | 0/11 | 0/16 | 0/14 | 0/14 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 0/2 | 0/4 | 0/11 | 0/16 | 0/14 | 0/14 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/40 | 0/43 | 0/2 | 0/4 | 0/11 | 0/16 | 0/14 | 0/14 | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT03535337/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT03535337/SAP_001.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT03535337/ICF_002.pdf